CLINICAL TRIAL: NCT00582322
Title: Genetic Studies in Breast Cancer
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Teresa Gilewski, MD, Memorial Sloan-Kettering Cancer Center
Other Study IDs: 92-007
Record Dates: First submitted 2007-12-21; First posted 2007-12-28 (Estimated); Last update posted 2009-07-20 (Estimated); Status verified 2009-07

CONDITIONS: Breast Cancer; Ovarian Cancer
Keywords: Breast Cancer; Ovarian Cancer; Family History; Genetic Studies
MeSH Terms: conditions — Breast Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood

SUMMARY:
The purpose of this study is to determine the specific genetic alterations associated with breast cancer. This will leat to a better understanding of the genetic causes of breast cancer.

DETAILED DESCRIPTION:
It is estimated that 175,000 new breast cancer cases and 44,5000 cancer deaths will result from female breast cancer in 1991. One of the most important risk factors is a family history of breast cancer. A susceptibility allele which accounts for a large proportion of familial breast cancer has been localized to chromosome 17q and attempts to clone the susceptibility are proceeding rapidly. The existence of recognized susceptibility loci and the awareness of a significan proportion of genetic predisposition and the associated penetrances remain unknown and are impossible to estimate without bias from previous studies. This study is designed to estimate heterogeniety and prenetrance in a series of unslected families, identify additional breast cancer susceptibility locs, as well as provide resources for gene isolation and mutation analysis studies.

ELIGIBILITY:
Inclusion Criteria:

* patient with breast cancer under age 41
* patient with bilateral breast cancer 41-50 years old or 41-50 years old with a first degree relative (mother, sister, daughter) with breast cancer diagnosed under age 50
* patient with ovarian cancer with first degree relative with either ovarian cancer diagnosed at any age or breast cancer diagnosed under age 60
* patient any age with either ovarian or breast cancer who have 2 first degree rleatives with either ovarian cancer diagnosed at any age or breast cancer diagnosed under age 50
* relatives of any of the above patients will be included in this trial if a genetic abnormality is found in the patient's blood sample

Exclusion Criteria:

N/A

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with breast cancer seen at MSKCC and healthy family members.
Sampling Method: Non-Probability Sample
Enrollment: 483 (Actual)
Dates: Start 1992-02; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Teresa Gilewski, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org